CLINICAL TRIAL: NCT04481230
Title: Assessment of 99mTc-NTP 15-5 Uptake on Cartilage, a New Proteoglycan Tracer: Phase I Clinical Trial
Brief Title: Assessment of 99mTc-NTP 15-5 Uptake on Cartilage, a New Proteoglycan Tracer
Acronym: CARSPECT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-000495-37
Record Dates: First submitted 2020-07-02; First posted 2020-07-22 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2023-09

CONDITIONS: Osteoarthritis, Knee; Breast Cancer
Keywords: cartilage; proteoglycan tracer
MeSH Terms: conditions — Osteoarthritis, Knee; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: dose escalation model
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 99mTc-NTP 15-5 (level 1) (Experimental): 99mTc-NTP 15-5 at a diagnostic activity of 5 MBq/kg
  Interventions: Drug: 99mTc-NTP 15-5 at a diagnostic activity of 5 MBq/kg
- 99mTc-NTP 15-5 (level 2) (Experimental): 99mTc-NTP 15-5 at a diagnostic activity of 10 MBq/kg
  Interventions: Drug: 99mTc-NTP 15-5 at a diagnostic activity of 10 MBq/kg
- 99mTc-NTP 15-5 (level 3) (Experimental): 99mTc-NTP 15-5 at a diagnostic activity of 15 MBq/kg
  Interventions: Drug: 99mTc-NTP 15-5 at a diagnostic activity of 15 MBq/kg

INTERVENTIONS:
Drug: 99mTc-NTP 15-5 at a diagnostic activity of 5 MBq/kg — 1 intravenous injection of 99mTc-NTP 15-5 at a diagnostic activity of 5 MBq/kg (D0)
  Arms: 99mTc-NTP 15-5 (level 1)
Drug: 99mTc-NTP 15-5 at a diagnostic activity of 10 MBq/kg — 1 intravenous injection of 99mTc-NTP 15-5 at a diagnostic activity of 10 MBq/kg (D0)
  Arms: 99mTc-NTP 15-5 (level 2)
Drug: 99mTc-NTP 15-5 at a diagnostic activity of 15 MBq/kg — 1 intravenous injection of 99mTc-NTP 15-5 at a diagnostic activity of 15 MBq/kg (D0)
  Arms: 99mTc-NTP 15-5 (level 3)

SUMMARY:
This study is a phase I clinical trial aimed to determine the recommended dose of 99mTc-NTP 15-5 to obtain the best tracer joints contrast on images without any toxicity.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria specific to group 1:

- Patient with painful unilateral osteoarthritis of the knee as femorotibial pattern defined by a radiographic score of 0/1 from Kellgren / Lawrence and an average WOMAC score> or equal to 4 and by minor disorders at MRI (MOCART 2.0 score> 70).

Inclusion criteria specific to group 2:

* Patient with non-metastatic breast cancer, hormone receptor positive, HER2 negative, with indication for adjuvant therapy with aromatase inhibitor; treatment not yet started.
* Age <60 years

Common inclusion criteria:

* Patient with at least 31 healthy joints (based on clinical assessment)
* signed written informed consent.
* Affiliation to a health insurance scheme.
* For women of childbearing age : negative serum pregnancy test at inclusion (less than 7 days prior injection of 99mTc-NTP 15-5).
* Willing and able to comply with study visits, treatment, exams and the protocol.

Exclusion Criteria:

* Patients <18 years of age.
* Pregnant or lactating patient.
* BMI> 30
* History of known allergy to excipients contained in the solution of 99mTc-NTP 15-5
* Chronic inflammatory rheumatism (rheumatoid arthritis, spondyloarthropathy, psoriatic arthritis, etc.) diffuse arthritis (at least 3 joints affected), autoimmune connectivitis, fibromyalgia.
* Known chronic joint pathology: osteoarthritis affecting at least 3 joints, autoimmune disease, inflammatory rheumatism (except unilateral knee arthritis).
* Persons deprived of their liberty, under guardianship / curatorship, or safeguard of justice.
* Treatment with NSAIDs or cessation of less than 48 h.
* Inability to comply with medical requirement / follow-up of the trial for geographic, family, social or psychological reasons. These conditions should be discussed with the patient before registration in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
determination of the recommended dose of 99mTc-NTP 15-5 to obtain the best tracer joints contrast on images without any toxicity | Imaging at Day 0 (30 minutes, 1 hour, 2 hours, 4 hours, 6 hours post-injection)
  defined as the dose from which 100% of patients will present a score 3 (semi-quantitative visual scale on whole body imaging) in at least 80% of healthy joints visualized on scintigraphies performed 2 h or less post-injection and without dose-limiting toxicity (DLT).
dose-limiting toxicity (DLT) | 1 week after injection of the 99mTc-NTP 15-5 (Day 0)
  defined as any grade 3-4 toxicity according to the NCI-CTCAE (version 4.03)

SECONDARY OUTCOMES:
3D quantification analysis | imaging at Day 0, 30 minutes, 2 hours, 4 hours, 6-8 hours after injection of the 99mTc-NTP 15-5
  TEMP Volumetric regions of interest (VOI) will be centered on cartilaginous zones, and on the corresponding bony diaphyses or vertebral body or the adjacent muscles. The articular uptake of 99mTc NTP-15-5 will thus be normalized to bone or muscle uptake.
Safety of 99mTc-NTP 15-5 (frequence of adverse events) | 1 week after injection of the 99mTc-NTP 15-5 (Day 0)
  according to the NCI-CTCAE (version 4.03)
Biodistribution of 99mTc-NTP 15-5 | imaging at Day 0, 30 minutes, 2 hours, 4 hours, 6-8 hours after injection of the 99mTc-NTP 15-5
  evaluated by measuring the percentage of injected activity of 99mTc-NTP 15-5 fixed on the target organs and on the pathological joints or healthy joints.
Pharmacokinetics of 99mTc-NTP 15-5 by assessment of Area Under the Curve (AUC) | at Day 0 during the first 8 hours after injection of the 99mTc-NTP 15-5
  radiation counting on whole blood and on plasma
Pharmacokinetics of 99mTc-NTP 15-5 by assessment of Maximum Concentration (Cmax) | at Day 0 during the first 8 hours after injection of the 99mTc-NTP 15-5
  radiation counting on whole blood and on plasma
Pharmacokinetics of 99mTc-NTP 15-5 by assessment of the time take to reach Cmax (Tmax) | at Day 0 during the first 8 hours after injection of the 99mTc-NTP 15-5
  radiation counting on whole blood and on plasma
Urinary elimination of 99mTc-NTP 15-5 | at Day 0 during the first 8 hours after injection of the 99mTc-NTP 15-5
  by counting
Dosimetry | imaging at Day 0, 30 minutes, 2 hours, 4 hours, 6-8 hours after injection of the 99mTc-NTP 15-5
  measurement of the absorbed dose per organ will be evaluated by quantitative analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Florent CACHIN, Pr, Principal Investigator — Centre Jean Perrin
Locations (2):
- France (2):
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU Clermont-Ferrand, Clermont-Ferrand

REFERENCES:
- [Derived] Chanchou M, Thivat E, Mathieu S, Levesque S, Sas N, Auzeloux P, Billoux T, Molnar I, Jouberton E, Rouanet J, Fois G, Maigne L, Penault-Llorca F, Miot-Noirault E, Durando X, Cachin F. [99mTc]Tc-NTP 15 - 5, a new proteoglycan tracer for functional imaging of joint cartilage: phase I (CARSPECT). EJNMMI Res. 2025 Sep 26;15(1):123. doi: 10.1186/s13550-025-01318-3. PMID 41003883
- [Derived] Thivat E, Chanchou M, Mathieu S, Levesque S, Billoux T, Auzeloux P, Sas N, Molnar I, Jouberton E, Rouanet J, Fois G, Maigne L, Galmier MJ, Penault-Llorca F, Miot-Noirault E, Durando X, Cachin F. Assessment of 99mTc-NTP 15-5 uptake on cartilage, a new proteoglycan tracer: Study protocol for a phase I trial (CARSPECT). Front Med (Lausanne). 2022 Oct 12;9:993151. doi: 10.3389/fmed.2022.993151. eCollection 2022. PMID 36314021